CLINICAL TRIAL: NCT04449796
Title: Predictive Value of Bio-impedance Vector Analysis on Long-term Outcome in ICU Patients
Status: Completed | Type: Observational
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Sponsor
Other Study IDs: nWMO 2018-312
Record Dates: First submitted 2020-06-24; First posted 2020-06-29 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-06

CONDITIONS: Long-term Outcome; Survival

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Phase angle, derived from bioimpedance analysis (BIA), reflects tissue quality and quantity in which cell mass, membrane integrity and hydration state are represented. Phase angle, as a measure of body composition, changes with the physical condition of patients and is associated with survival in several disease states and during ICU admission. Aim of the study is to explore the predictive value of the phase angle for long term ICU outcome.

DETAILED DESCRIPTION:
Phase angle, derived from bioimpedance analysis (BIA), reflects tissue quality and quantity in which cell mass, membrane integrity and hydration state are represented. Phase angle, as a measure of body composition, changes with the physical condition of patients and is associated with survival in several disease states and during ICU admission. Aim of the study is to explore the predictive value of the phase angle for long term ICU survival.

A single-centre prospective observational cohort will be performed with consecutive patients, elective and non elective, admitted to the ICU between 1st June 2018 and 1st June 2019. Demographic data, APACHE III, comorbidity and phase angle are collected and the ICU- , hospital- and 6 months survival will be registered.

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted to the ICU, elective and acute.

Exclusion Criteria:

* age below 18
* Length of stay at ICU < 6 hours
* All invalid bio-impedence analysis (BIA) measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patiens admitted to the ICU
Sampling Method: Probability Sample
Enrollment: 1025 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
3 months survival | 3 months
  100% minus all-cause mortality at three month post ICU
6 months survival | 6 months
  100% minus all-cause mortality at six month post ICU
12 months survival | 12 months
  100% minus all-cause mortalityat twelve month post ICU

CONTACTS AND LOCATIONS:
Overall Officials: E.C. Boerma, MD PhD, Principal Investigator — Frisius Medisch Centrum
Locations (1):
- Medical Centre Leeuwarden - Intensive Care Unit, Leeuwarden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stellingwerf F, Beumeler LFE, Rijnhart-de Jong H, Boerma EC, Buter H. The predictive value of phase angle on long-term outcome after ICU admission. Clin Nutr. 2022 Jun;41(6):1256-1259. doi: 10.1016/j.clnu.2022.03.029. Epub 2022 Apr 6. PMID 35504168